CLINICAL TRIAL: NCT06436534
Title: A Randomized, Double-blind, Placebo-controlled, Single-center Clinical Trial of Ganciclovir Capsules in the Treatment of Refractory Moderate-to-severe Allergic Rhinitis
Brief Title: Efficacy and Safety of Ganciclovir Capsules in the Treatment of Refractory Moderate-to-severe Allergic Rhinitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chen Jianjun, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENTAR-GCV20240205
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Ganciclovir; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ganciclovir (Experimental): Screening phase(Day -14±2~0):Mometasone furoate nasal spray(50μg/spray), take 1 spray once a day.
  Treatment phase(Day 1~14±2): Ganciclovir capsules(250mg), take 2 capsules twice a day + Mometasone furoate nasal spray(50μg/spray), take 1 spray once a day.
  Follw-up phase(Day 14~28±2):Mometasone furoate nasal spray(50μg/spray), take 1 spray once a day.
  Interventions: Drug: Ganciclovir Oral Capsule; Drug: Mometasone Nasal
- Placebo (Placebo Comparator): Screening phase(Day -14±2~0):Mometasone furoate nasal spray(50μg/spray), take 1 spray once a day.
  Treatment phase(Day 1~14±2): Ganciclovir simulant capsules(0mg), take 2 capsules twice a day + Mometasone furoate nasal spray(50μg/spray), take 1 spray once a day.
  Follw-up phase(Day 14~28±2):Mometasone furoate nasal spray(50μg/spray), take 1 spray once a day.
  Interventions: Drug: Ganciclovir Simulant Oral Capsule; Drug: Mometasone Nasal

INTERVENTIONS:
Drug: Ganciclovir Oral Capsule — 2-week treatment phase：Ganciclovir capsules(250mg), take 2 capsules twice a day
  Other Names: Ganciclovir
  Arms: Ganciclovir
Drug: Ganciclovir Simulant Oral Capsule — 2-week treatment phase：Ganciclovir simulant capsules(0mg), take 2 capsules twice a day
  Other Names: Ganciclovir
  Arms: Placebo
Drug: Mometasone Nasal — From screening phase to follow-up phase：Mometasone furoate aqueous nasal spray(50μg/spray), take 1 spray once a day
  Other Names: Mometasone furoate aqueous nasal spray; NASONEX; Mometasone furoate nasal spray

SUMMARY:
The goal of this clinical trial is to learn about the clinical efficacy and safety of ganciclovir (GCV) capsules in the treatment of refractory moderate-to-severe allergic rhinitis. The main questions it aims to answer are:

1. Whether ganciclovir improve nasal symptoms and life quality in patients with refractory moderate-to-severe allergic rhinitis.
2. Whether ganciclovir is safe for the treatment of allergic rhinitis.

Participants with refractory moderate-to-severe allergic rhinitis will be included in the trial based on the inclusion and exclusion criteria, and randomized into experimental and control groups.

The two groups will be treated with blinded ganciclovir capsules or placebo for two weeks, with the background therapy of mometasone furoate aqueous nasal spray. A placebo is a look-alike capsule that contains no active drug. Nasal symptom scores, nasal secretions, blood samples and adverse events will be collected during the visits.

Researchers will compare the experimental and control groups to see whether ganciclovir improve symptoms and is safe for the treatment of refractory moderate-to-severe allergic rhinitis.

DETAILED DESCRIPTION:
Ganciclovir (GCV) is clinically used for the treatment of DNA viral infections. In clinical practice, we have found that patients with refractory AR have improved nasal symptoms after oral administration of ganciclovir. In clinical practice, we have found that patients with refractory AR have improved nasal symptoms after oral administration of ganciclovir. To further explore the role of GCV in the treatment of refractory allergic rhinitis, we have conducted an interventional non-randomised cohort study of GCV for refractory AR. The results found that 65% of all refractory AR patients included in the observation were effectively treated with GCV. Based on the previous discovery in the clinical practice, the conjecture is proposed that ganciclovir may improve symptoms in allergic rhinitis patients, in particular the patients with refractory moderate-to-severe allergic rhinitis. Thus, the randomized, double-blind, placebo-controlled clinical trial was designed to explore the validity of this hypothesis.

The research involves three phases: screening phase(Day-14±2~0)；baseline (Day1)；treatment phase (Day1~14)；follow-up phase (Day14~28).

In the screening phase, anterior rhinoscopy, serum specific IgE test, skin prick test, total nasal symptom scores (TNSS), visual analogue scale (VAS) scores, Allergic Rhinitis Control Test (ARCT) score will be performed for participants. Participants who meet the inclusion and exclusion criteria will enter the treatment phase and receive the medication for two weeks. At the end of the treatment, researchers will follow participants for two weeks to track efficacy and safety.

Researchers will collect participants' symptom scores, nasal secretions and blood. The biological specimens will be used to test for indicators that support the determination of therapeutic efficacy. Vital signs, blood routine examination, urine routines, liver function test, kidney function test and electrocardiograms will be measured for participants before and after treatment to assess the safety of ganciclovir.

The data collected will be statistically analyzed to examine the clinical efficacy and safety of ganciclovir capsules in the treatment of refractory moderate-to-severe allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years.
2. Diagnosed with moderate-to-severe perennial allergic rhinitis based on Chinese guideline for diagnosis and treatment of allergic rhinitis (2022, revision) with Allergic Rhinitis Control Test (ARCT) score <20.
3. Total Nasal Symptom Score (TNSS) ≥6 or at least two of the four subdomains(sneezing, rhinorrhea, nasal itching, and nasal obstruction) ≥2 at the time of both screening and randomization. And the improvement in TNSS was assessed as < 30% at randomization compared to screening.
4. The participant is allergic to dust mites or other perennial allergens
5. Voluntarily participate in the clinical trial and sign the informed consent.

Exclusion Criteria:

1. Participants with hypersensitivity to ganciclovir capsules and its excipients.
2. Have symptoms of viral infection, fever and other systemic symptoms in the past 2 weeks.
3. Pregnant or lactating women and participants who have pregnancy plan during the study period.
4. Participants with severe neutropenia (absolute neutrophil count less than 0.5*10^9/L) or severe thrombocytopenia (platelet count less than 2.5*10^10/L).
5. Comorbidities such as upper and lower respiratory tract infections, history of acute or chronic sinusitis, dry rhinitis, atrophic rhinitis, severe deviated septum and asthma.
6. Participants with other severe heart, lung, liver and kidney disease.
7. Participants who had received any live or attenuated vaccine within 4 weeks prior to baseline or intended to receive live or attenuated vaccine (or BCG treatment) during the study period or within 4 weeks after the last administration of the investigational drug product.
8. Participants with a history of HIV infection or who test positive for HIV serology.
9. Participants currently infected or chronically infected with hepatitis B virus (HBV) or hepatitis C virus (HCV).
10. Participants with cirrhosis and/or chronic hepatitis.
11. Participants who have been diagnosed with active parasitic infections or are at high risk of developing such infections.。
12. Participants with a known or suspected history of immunosuppression, including a history of invasive opportunistic infections (e.g., histoplasmosis, listeriosis, coccidioidomycosis, pneumosporidiosis, aspergillosis). Or participants with what researchers believe to be unusually frequent, recurring, or prolonged infections.
13. Participants with a known history of malignancy within 5 years prior to screening.
14. Participants with severe co-morbidities that, in the opinion of the investigator, would adversely affect their participation in this study.
15. Participants with combined neurological or psychiatric disorders who are unable or reluctant to cooperate.
16. Participants with disabilities prescribed by law (blind, deaf, mute, mentally challenged, mentally handicapped, etc.).
17. Participants suspected or having a history of alcohol and drug abuse.
18. Other participants who have been involved in other clinical trials within 3 months before the screening.
19. The researchers consider it inappropriate to participate in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of improvement in TNSS scores | From baseline to the end of treatment phase(2 weeks)
  After 2 weeks of treatment phase, the investigator assess the rate of change in the difference in TNSS from baseline. Calculated as (total post-treatment symptom score - total pre-treatment symptom score)/total pre-treatment symptom score × 100%.

SECONDARY OUTCOMES:
Total effective rate | From baseline to the end of treatment phase(2 weeks)
  Participants with a >30% decrease in total nasal symptom scores (TNSS) after 2 weeks of treatment are considered effective. The percentage of participants effective on treatment will be assessed as total effective rate.
Rate and absolute value of change in TNSS and four subdomains. | From baseline to the end of treatment phase(2 weeks)
  TNSS assesses symptom severity in four subdomains consisting of sneezing, rhinorrhea, nasal itching, and nasal obstruction. Each subdomain is rated on a scale of 0 (no symptoms) to 3 (severe symptoms that are difficult to tolerate and interfere with daily activity). The overall TNSS score is the sum of all four symptoms resulting in a maximum score of 12.
  After the treatment phase, evaluate the rate and absolute value of change in TNSS and four subdomains from baseline.
Rate and absolute value of change in visual analogue scale (VAS) scores. | From baseline to the end of treatment (2 weeks)
  The VAS ranges from 0 to 100. A score of 0 corresponds to no symptoms and 100 corresponds to the worst symptoms.
  After the treatment phase, evaluate the rate and absolute value of change in VAS scores from baseline.
Rate and absolute value of change in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | From baseline to the end of treatment (2 weeks)
  RQLQ is a validated QOL instrument consisting of 28 questions in seven domains (limited activity, sleep, practical problems, nasal symptoms, eye symptoms, emotional function, and non-nose/eye or other symptoms). Each domain is graded from zero (not impaired at all) to six (severely impaired), and the overall RQLQ is the mean score of all 28 responses.
  After the treatment phase, evaluate the rate and absolute value of change in RQLQ scores from baseline.
Change in mean TNSS during a 2-week administration period | During the 2-week administration period
  Participants assess the TNSS score on a daily basis. TNSS assesses symptom severity in four subdomains consisting of sneezing, rhinorrhea, nasal itching, and nasal obstruction. Each subdomain is rated on a scale of 0 (no symptoms) to 3 (severe symptoms that are difficult to tolerate and interfere with daily activity). The overall TNSS score is the sum of all four symptoms resulting in a maximum score of 12.
  After the treatment phase, evaluate the change in mean TNSS during a 2-week administration period from baseline.
Rate and absolute value of change in TNSSand four subdomains, VAS, RQLQ scores in follow-up phase | From baseline to the end of follow-up phase (4 weeks)
  After the follow-up phase, evaluate the rate and absolute value of change in TNSS, VAS, RQLQ scores from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Chen, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demoly P, Jankowski R, Chassany O, Bessah Y, Allaert FA. Validation of a self-questionnaire for assessing the control of allergic rhinitis. Clin Exp Allergy. 2011 Jun;41(6):860-8. doi: 10.1111/j.1365-2222.2011.03734.x. Epub 2011 Apr 25. PMID 21518040
- [Background] Mathur V, Burai R, Vest RT, Bonanno LN, Lehallier B, Zardeneta ME, Mistry KN, Do D, Marsh SE, Abud EM, Blurton-Jones M, Li L, Lashuel HA, Wyss-Coray T. Activation of the STING-Dependent Type I Interferon Response Reduces Microglial Reactivity and Neuroinflammation. Neuron. 2017 Dec 20;96(6):1290-1302.e6. doi: 10.1016/j.neuron.2017.11.032. PMID 29268096
- [Background] Ding Z, Mathur V, Ho PP, James ML, Lucin KM, Hoehne A, Alabsi H, Gambhir SS, Steinman L, Luo J, Wyss-Coray T. Antiviral drug ganciclovir is a potent inhibitor of microglial proliferation and neuroinflammation. J Exp Med. 2014 Feb 10;211(2):189-98. doi: 10.1084/jem.20120696. Epub 2014 Feb 3. PMID 24493798
- [Background] Crumpacker CS. Ganciclovir. N Engl J Med. 1996 Sep 5;335(10):721-9. doi: 10.1056/NEJM199609053351007. No abstract available. PMID 8786764
- [Background] Demoly P, Calderon MA, Casale T, Scadding G, Annesi-Maesano I, Braun JJ, Delaisi B, Haddad T, Malard O, Trebuchon F, Serrano E. Assessment of disease control in allergic rhinitis. Clin Transl Allergy. 2013 Feb 18;3(1):7. doi: 10.1186/2045-7022-3-7. PMID 23419058